CLINICAL TRIAL: NCT04701437
Title: HCV-ACCELERATE Advanced Care Coordination and Enhanced Linkage and Retention Among Transitional Re-Entrants
Brief Title: Advanced Care Coordination and Enhanced Linkage and Retention Among Transitional Re-Entrants
Acronym: ACCELERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Prisma Health-Upstate (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-12458; 4R00DA043011 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2021-01-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C
Keywords: recently incarcerated; Hepatitis C; peer mentor
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-enhanced intervention (Experimental): Those randomized to the peer-enhanced intervention group will be contacted by a peer mentor within 72 hours of enrollment to discuss the early release period, readiness for HCV treatment, and identify ancillary needs. Individuals randomized to this arm will be provided a study cell phone.
  Interventions: Behavioral: Peer mentor
- Standard of care (Placebo Comparator): If randomized to the standard of care intervention, the participant will only receive passive referral to HCV-care.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Peer mentor — Peer mentors will contact participants within 72 hours of enrollment to discuss the early release period, gauge their readiness for HCV treatment, and identify ancillary needs. They will also accompany the participant to their first medical appointment with an HCV provider and any future appointments if requested by the participant. Peer mentors will offer participants social support throughout the 6 months they are enrolled in the study.
  Arms: Peer-enhanced intervention
Behavioral: Standard of care — Passive referral to a HCV provider
  Arms: Standard of care

SUMMARY:
The overarching goal of this study is to develop a peer-based care coordination intervention for individuals with Hepatitis C Virus (HCV) who were recently released from correctional settings to promote linkage to and retention in HCV care. The investigators will assess the existing barriers and facilitators of HCV treatment initiation, HCV treatment completion, and sustained virologic response among individuals recently released from a U.S. jail or prisons in a randomized control trial. This study will assess the feasibility and process measures of a peer-enhanced HCV care coordination intervention among recently incarcerated individuals.

DETAILED DESCRIPTION:
The proposed 2-year study will be a block stratified, randomized controlled trial. Once consented and enrolled, participants will be randomly assigned to either the peer-enhanced intervention or referred to standard clinical care. The investigators will enroll 80 former inmates with chronic HCV who have been released from incarceration within the past 6 months. It is expected that enrollment will be completed by the fourth quarter of the first year. This will allow sufficient time for HCV treatment uptake, completion, determination of Sustained Virologic Response (SVR), and assessment of reinfection. Individual participant follow-up will be 3 months on average for treatment, 3 months for SVR, and 3 months to assess for reinfection.

Elucidating the barriers and facilitators in the re-entry care cascade (as well as how they may be overcome) will be critical in designing sustainable models of care for HCV-infected former inmates. The investigators hypothesize that a peer-enhanced strategy will be more effective than standard referral in improving linkage to, and retention in, HCV care among individuals recently released from correctional settings.

ELIGIBILITY:
Inclusion Criteria:

* currently incarcerated or recently released from a U.S. jail or prison (6 months)
* Chronic HCV with documented detectable viral load
* 18 years old
* Fluent in English or Spanish
* Resident of the Upstate area of South Carolina

Exclusion Criteria:

* Unable to sign informed consent
* Life expectancy of less than 1 year
* Plans to relocate from the Upstate area of South Carolina in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Linkage to care | 6 months
  A visit with an HCV treatment provider

SECONDARY OUTCOMES:
HCV treatment initiation | up to 3 months after linkage to care
  Initiating HCV treatment and the number of days following release from the correctional setting to initiation of HCV treatment
Treatment completion | up to 3 months after treatment initiation
  Completing HCV treatment, as determined by EMR
HCV cure | 3 months after treatment completion
  Achieving HCV cure, as determined by EMR
Reinfection | 12 months after treatment completion
  Determined by EMR

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Akiyama, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine; Alain Litwin, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Prisma Health-Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riback LR, Davis M, King A, Boswell K, Moore C, Dendy B, Hoeflich C, Heo M, Litwin AH, Akiyama MJ. Rationale, design, and methodology of a randomized controlled trial evaluating the impact of peer-enhanced care coordination on linkage to HCV care among formerly incarcerated individuals. Contemp Clin Trials. 2025 Dec;159:108137. doi: 10.1016/j.cct.2025.108137. Epub 2025 Nov 3. PMID 41192754